CLINICAL TRIAL: NCT00665379
Title: Prospective, Randomized Controlled Trial Comparing the Effect of 3M Coban 2 Layer Compression System Versus Trico Bandages in the Treatment of Leg Lymphedema.
Brief Title: Comparative Trial in Compression Therapy in Leg Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, R.J. Damstra, MD PhD, Nij Smellinghe Hosptial
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS1NL
Record Dates: First submitted 2008-04-17; First posted 2008-04-23 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Leg Lymphedema
Keywords: leg lymphedema; volume measurement; compression therapy; interface pressure; static stiffness index (SSI); volume change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Regular compression therapy with non elastic trico bandaging
  Interventions: Other: Regular Compression therapy (Trico bandages)
- 2 (Active Comparator): New two layer compression bandage coban 2
  Interventions: Other: New Compression therapy (C2L bandages)

INTERVENTIONS:
Other: Regular Compression therapy (Trico bandages) — Application of marketed Trico compression bandages used for treatment by trained specialists with assessment of the subbandage pressure and volume reduction. The bandages are applicated in patients with leg lymphedema at t=0 hour, t=2 hours. Comparison is made at t=2 hours, t= 24 hours
  Other Names: trico bandages
  Arms: 1
Other: New Compression therapy (C2L bandages) — Application of marketed compression bandages C2L used for treatment by trained specialists with assessment of the subbandage pressure and volume reduction. he bandages are applicated in patients with leg lymphedema at t=0 hour, t=2 hours. Comparison is made at t=2 hours, t= 24 hours
  Other Names: coban 2
  Arms: 2

SUMMARY:
The purpose of this trial is to study the effect of the 3M Coban 2 Layer Compression System (hereafter C2L) in the treatment of leg lymphedema compared to the traditional treatment with Trico bandages.

DETAILED DESCRIPTION:
The goal of this prospective, randomized, controlled trial with CE marked product is to study the effectiveness (volume reduction) of 24-hour compression therapy for lymphedema, comparing C2L and Trico bandaging. Therefore 30 patients with leg lymphedema are included.

Application of marketed compression bandages (C2L or Trico bandages) used for treatment by trained specialists with assessment of the subbandage pressure and volume reduction.

Measurements are carried out at:

Volumetry:

Measurements after 0h, 2h and 24 h by using classic water displacement apparatus.

Pressure:

Measurements after 0h, 2h (pre and post bandage change) and 24 h;

* supine and standing to calculate the SSI;
* supine with and without dorsal flexion.

for the pressure measurement a Kikuhime (large pads) dice is used. At each new bandaging to document the SSI and the effect of dorsiflexion in the supine position

* The subbandage pressure is measured on the medial aspect of the lower leg at the transition of the gastrocnemius muscle into the Achilles' tendon (B1) (Partsch H. et al. Dermatol Surg 2006; 32: 224-233).
* Fix the sensor (sensor and tube sheathed with Cellona Soft Padding)

Statistical analysis; Analysis of variance (ANOVA) comparing volume, supine subbandage pressure with and without dorsiflexion, and SSI for the used bandages

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* More than 18 years of age
* Patients with distal lymphedema of the leg requiring multilayer lymphedema bandaging of the leg
* The patient is able to understand the study and is willing to give written informed consent to the study

Exclusion Criteria:

* Allergy against one of the used materials
* Proximal lymphedema (involvement of thigh, genitalia)
* Severe systemic diseases causing peripheral oedema
* Acute superficial or deep vein thrombosis
* Arterial occlusive disease (stadium II, III or IV) or arm/leg blood pressure index (ALPI)<0,8
* Local infection in the therapy area
* Auto-immunological disorders or vasculitis
* Use of systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
volume decrease in relation to interface pressure after application of two types of bandages. | enrollment of 30 patients

SECONDARY OUTCOMES:
Pressure drop after 2 hours and 24 hours of bandaging | after application, at 2 hours and 24 hours after application of bandage

CONTACTS AND LOCATIONS:
Overall Officials: RJ Damstra, MD, Principal Investigator — Nij Smellinghe Hospital; H Partsch, PhD, Study Director — Private practice, wien
Locations (1):
- Nij Smellinghe hospital, Drachten, Provincie Friesland, Netherlands